CLINICAL TRIAL: NCT00265031
Title: HD12 for Advanced Stages
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Cologne (Other)
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: HD12
Record Dates: First submitted 2005-12-12; First posted 2005-12-13 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2007-08

CONDITIONS: Hodgkin´s Lymphoma
Keywords: Hodgkin´s Lymphoma; advanced stages
MeSH Terms: interventions — Cyclophosphamide; Doxorubicin; Etoposide; Procarbazine; Prednisone; Vincristine; Bleomycin; Radiotherapy

INTERVENTIONS:
Drug: Cyclophosphamide
Drug: Adriamycin
Drug: Etoposide
Drug: Procarbazine
Drug: Prednisone
Drug: Vincristine
Drug: Bleomycin
Procedure: radiation therapy

SUMMARY:
This study is designed to test (1) whether the BEACOPP dosage can be reduced to baseline in the last 4 cycles without loss of effectiveness, and (2) whether consolidating irradiation is necessary following effective chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

* Hodgkin´s lymphoma (histologically proven)
* CS(PS) IIB with one or both of the risk factors:

  1. bulky mediastinal mass (> 1/3 of maximum transverse thorax diameter)
  2. extranodal involvement
* CS(PS) III, IV
* written informaed consent

Exclusion Criteria:

* Leukocytes <3000/microl
* Platelets <100000/microl
* Hodgkin´s Disease as "composite lymphoma"
* Activity index (WHO) < grade 2

Ages: 16 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Volker Diehl, Prof., Principal Investigator — University of Cologne

REFERENCES:
- [Result] Borchmann P, Haverkamp H, Diehl V, Cerny T, Markova J, Ho AD, Eich HT, Mueller-Hermelink HK, Kanz L, Greil R, Rank A, Paulus U, Smardova L, Huber C, Dorken B, Nerl C, Krause SW, Mueller RP, Fuchs M, Engert A. Eight cycles of escalated-dose BEACOPP compared with four cycles of escalated-dose BEACOPP followed by four cycles of baseline-dose BEACOPP with or without radiotherapy in patients with advanced-stage hodgkin's lymphoma: final analysis of the HD12 trial of the German Hodgkin Study Group. J Clin Oncol. 2011 Nov 10;29(32):4234-42. doi: 10.1200/JCO.2010.33.9549. Epub 2011 Oct 11. PMID 21990399
- [Derived] von Tresckow B, Kreissl S, Goergen H, Brockelmann PJ, Pabst T, Fridrik M, Rummel M, Jung W, Thiemer J, Sasse S, Burkle C, Baues C, Diehl V, Engert A, Borchmann P; German Hodgkin Study Group. Intensive treatment strategies in advanced-stage Hodgkin's lymphoma (HD9 and HD12): analysis of long-term survival in two randomised trials. Lancet Haematol. 2018 Oct;5(10):e462-e473. doi: 10.1016/S2352-3026(18)30140-6. PMID 30290903
- See also: Description of study i German (Website of the Competence Network Malignant Lymphoma) — http://www.lymphome.de/Gruppen/GHSG/